CLINICAL TRIAL: NCT06595563
Title: HER2 Molecular Imaging With 89Zr-trastuzumab PET/CT as a Predictive Biomarker for Antibody-drug Conjugate Sequencing in Patients With Advanced HER2-positive Breast Cancer
Acronym: ZEPHIR-02
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IJB-ZEPHIR02-2024
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2024-09

CONDITIONS: HER2-positive Metastatic Breast Cancer; HER2-positive Advanced Breast Cancer
MeSH Terms: interventions — Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HER2 PET/CT "positive" (Experimental): Subjects classified as HER2-PET/CT positive (cohort A) will receive T-DM1, IV 3.6mg/kg every 3 weeks, as monotherapy. HER2-PET/CT positive pattern: The entire or majority of the tumour load shows significant tracer uptake.
  Interventions: Drug: Trastuzumab emtansine
- HER2 PET/CT "negative" (No Intervention): Subjects classified as HER2 PET/CT negative (cohort B) will receive treatment of physician's choice (TPC) as per the best local clinical practice. Subsequent treatment will be collected and the subject will enter survival follow-up. HER2-PET/CT negative pattern: The dominant part or all of the tumour load lacks significant tracer uptake.

INTERVENTIONS:
Drug: Trastuzumab emtansine — T-DM1 will be administered IV at a dose of 3.6 mg/kg every 3 weeks. (21 days +/- 3 days) until disease progression, unacceptable toxicity or request of the subject to withdraw from the study. The total dose will depend on the subject's weight on day 1 of each T-DM1 cycle.
  Other Names: T-DM1
  Arms: HER2 PET/CT "positive"

SUMMARY:
ZEPHIR-02 is a multicentre, open-label phase II study that will enroll subjects with HER2-positive advanced/metastatic breast cancer (mBC) who have experienced disease progression under trastuzumab deruxtecan (T-DXd) in the metastatic setting.

All subjects will undergo baseline biopsy, blood collection, FDG-PET/CT and 89Zr-trastuzumab PET/CT (HER2-PET/CT) and will be classified as HER2-PET/CT positive or negative, as previously described in the ZEPHIR trial. Subjects classified as "positive" (cohort A) will receive T-DM1 as monotherapy, IV 3.6mg/kg every 3 weeks (21 days +- 3 days) until disease progression, unacceptable toxicity or request of the subject to withdraw from the study. Early FDG PET/CT will be performed before cycle 2 of T-DM1 to assess the response to the treatment. Routine tumour assessments will be performed with FDG-PET/CT until efficacy follow-up is completed. After 2 years of treatment with T-DM1 received by the subject, physician can consider to space the cycles up to 6 weeks.

Subjects classified as HER2-PET/CT negative (cohort B) will receive treatment of physician's choice as per the best local clinical practice.

The study also includes mandatory translational procedures (i.e. collection of tumour biopsy during pre-treatment period and blood samples at pre-specified time points) for exploratory molecular analyses.

DETAILED DESCRIPTION:
ZEPHIR-02 is a multicentre, open-label phase II study that will enroll subjects with HER2-positive advanced/metastatic breast cancer (mBC) who have experienced disease progression under trastuzumab deruxtecan (T-DXd) in the metastatic setting.

All subjects will undergo baseline biopsy, blood collection, FDG-PET/CT and 89Zr-trastuzumab PET/CT (HER2-PET/CT) and will be classified as HER2-PET/CT positive or negative, as previously described in the ZEPHIR trial. Focusing on a central visual "patient-based" classification that captures the entire disease burden, a side-by-side display will be used, comparing baseline FDG-PET/CT (which identifies all FDG-positive metastases regardless of their HER2-imaging status) and HER2-PET/CT. Subjects will be categorized into two HER2-PET/CT patterns (positive vs. negative) based on proportion of FDG-avid tumour load with significant 89Zr-trastuzumab uptake. Lesion uptake will be considered significant/pertinent if it is visually higher than the local background.

* HER2-PET/CT positive pattern: The entire or majority of the tumour load shows significant tracer uptake.
* HER2-PET/CT negative pattern: The dominant part or all of the tumour load lacks significant tracer uptake.

Subjects classified as "positive" (cohort A) will receive T-DM1 as monotherapy, IV 3.6mg/kg every 3 weeks (21 days +- 3 days) until disease progression, unacceptable toxicity or request of the subject to withdraw from the study. FDG-PET/CT will be performed before cycle 2 of T-DM1 for early assessment of response and then again before cycle 4. At the early FDG-PET/CT assessment (before cycle 2), response assessment will be done using a cut-off of 15% based on the CONSIST criteria. Subjects who demonstrate a partial or complete response (responders) and will continue treatment with T-DM1. Subjects who exhibit stable disease or disease progression (non-responders) will discontinue study treatment and enter the survival follow-up period. For responders, subsequent metabolic evaluations will be performed every 3 months, with FDG-PET/CT. Treatment response will be assessed according to metabolic response. For these subjects, blood samples will be obtained at all metabolic reassessments (mandatory).

The subjects with HER2 PET/CT classified as "negative" (cohort B) will receive treatment of physician's choice (TPC) as per the best local clinical practice. Subsequent treatment will be collected and the subject will enter survival follow-up.

All enrolled subjects will undergo a mandatory biopsy during the pre-treatment period. Of note, results of DNA sequencing on the biopsy will be communicated to the treating oncologist, to potentially inform post progression therapy.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status ≤ 1
* Must have histologically or cytologically confirmed progressive advanced/metastatic HER2-positive breast carcinoma as per the updated American Society of Clinical Oncology (ASCO) - College of American Pathologists (CAP) guidelines according to local testing. HER2 status may be determined in the primary breast cancer tumour or, when not available, in a metastatic lesion.
* Multifocal unilateral or bilateral breast adenocarcinoma tumours are allowed if all tested HER2-positive, according to local testing
* Prior treatment with taxane, trastuzumab and pertuzumab (early or advanced setting) and T-DXd (metastatic setting). In order to be eligible, patients subjects must have received T-DXd as the last systemic metastatic treatment line before inclusion, and presented disease progression on this drug.

Prior therapy with tucatinib, trastuzumab, and capecitabine, in advanced setting, is permissible, provided that T-DXd serves as the last systemic metastatic treatment line before inclusion, and patient subject presented disease progression on this drug.

* Life expectancy ≥ 6 months.
* At screening FDG-PET at least two "target" lesions are required to fulfil the following criteria: (1) anatomically transaxial diameter ≥ 1.5 cm and (2) metabolically assessable with a maximum standard uptake value corrected for lean body mass (SUVmax) ≥ 1.5 x SUVmean + 2 standard deviations (SD) of the liver measured in a 3-cm-diameter spherical volume of interest (VOI) in normal liver parenchyma.

In case of suspected liver metastasis, a lesion should have a SUVmax ≥ 2 x SUVmean + 3 SD of the blood pool measured in a 1 cm-diameter VOI within descending thoracic aorta. Lesions pre-treated with irradiation are not eligible for consideration as "target" lesions.

* Adequate Bone Marrow Function including:

  * Absolute Neutrophil Count (ANC) ≥1000/μL or ≥1x109/L.
  * Platelets ≥100,000/μL or ≥ 100 x 109/L.
  * Haemoglobin ≥ 9 g/dL.
* Adequate Renal Function including serum creatinine ≤ 1.5 x upper limit of normal (ULN) or estimated creatinine clearance ≥ 60 ml/min as calculated using the method standard for the institution.
* Adequate Liver Function, including all the following parameters:

  * Total serum bilirubin ≤ 1.5 x ULN unless the patient subject has documented Gilbert syndrome.
  * Aspartate and Alanine Aminotransferase (AST and ALT) ≤ 2.5x ULN.
* Current left ventricular ejection fraction (LVEF) ≥ 50% on echocardiography or multiple-gated acquisition scanning and no history of a LVEF < 40% or symptomatic heart failure or a recent myocardial infarction.
* Willingness to provide tumour tissue (mandatory biopsy) and blood samples (mandatory) for translational research activities.
* Willingness to comply with the protocol for the duration of the study including treatment and scheduled visits and examinations.
* Signed Informed Consent form (ICF) obtained prior to any study related procedure.

Inclusion criterion applicable to FRANCE only:

* Affiliated to the French Social Security System

Exclusion Criteria:

* Prior exposure to T-DM1 for the treatment of metastatic BC. For subjects exposed to T-DM1 for the treatment of early BC, subjects must not have relapsed while on or within 12 months of finishing treatment with T-DM1.
* Brain metastasis as sole metastasis and/or symptomatic or requiring therapy to control symptoms.
* History of interstitial lung disease / pneumonitis (grade 3 or 4) during the prior treatment with T-DXd.
* Cardiopulmonary dysfunction as defined by any of the following:

  * Significant symptoms (Grade ≥ 2) relating to LV dysfunction, cardiac arrhythmia, or cardiac ischemia while or since receiving preoperative therapy.
  * Uncontrolled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg)
  * Inadequately controlled angina, serious cardiac arrhythmia not controlled by adequate medication, severe conduction abnormality, or clinically significant valvular disease
  * Screening LVEF < 50% by either ECHO or MUGA
  * History of NCI CTCAE (Version 4.0) Grade ≥ 3 symptomatic congestive heart failure (CHF) or New York Heart Association (NYHA) criteria Class ≥ II
  * History of a decrease in LVEF to < 40% or symptomatic CHF with prior trastuzumab treatment (e.g., during preoperative therapy)
  * Myocardial infarction within 12 months prior to randomization
  * Requirement for continuous oxygen therapy
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to trastuzumab or excipients.
* Contra-indication for treatment with T-DM1.
* The number of subjects included in this trial, considered as "rapid progressors" (Rapid progressors defined as progressive disease within the first 6 months of T-DXd therapy) will be capped at 10% at enrolment (no more than 7 subjects out the 78 subjects planned to be recruited). After the first 7 "rapid progressors" included, progression within the first 6 months of T-DXd therapy will be considered as an exclusion criterion.
* Any known liver disease, including known carriers of hepatitis B virus, hepatitis C, autoimmune hepatic disorders and sclerosing cholangitis.
* Concurrent, serious, uncontrolled infections or known infection with HIV. Prior history of other invasive cancer in the past 5 years except basal or squamous cell carcinoma of skin that has been definitively treated.
* Pregnant and/or lactating women, or intending to become pregnant during the study. Serum pregnancy test (for subjects of childbearing potential) positive within 15 days prior to enrolment.
* Women of childbearing potential refusing to use one highly effective method of contraception from ICF signature, during the course of the study and at least 7 months after the last administration of T-DM1.
* Men with childbearing potential partner refusing to use condom during the course of this study and for at least 7 months after the last administration of T-DM1.
* Subject with a significant medical, neuro-psychiatric, or surgical condition, currently uncontrolled by treatment, which, in the principal investigator's opinion, may interfere with completion of the study.

Exclusion criterion applicable to FRANCE only:

* Vulnerable persons according to the article L.1121-6 of the Public Health Code, adults who are the subject of a measure of legal protection or unable to express their consent according to article L.1121-8 of the Public Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Characterization of genomic alterations and HER2 expression (cohorts A and B). | Through study completion, up to 2 years depending on the cohort
  To characterize the tumour landscape (molecular alterations on tissue and HER2 expression and its heterogeneity) in HER2-positive mBC (cohorts A and B) after at least 1 line of systemic therapy for advanced disease in order to better inform the oncologist and the subject regarding next treatment options.
Time to treatment failure (TTF) | During study treatment period (from C1 of T-DM1 until discontinuation), up to 1 year on average
  The time to treatment failure (TTF), defined as the time from T-DM1 start to discontinuation for any reason, including disease progression (clinical or image-based on 18FDG-PET/CT), treatment toxicity or death in participants included in cohort A (per metabolic response).
  Time to Treatment Failure (TTF) of subjects in cohort A and its survival probability measures (median survival, survival rate at month 6) will be estimated using Kaplan-Meier method

SECONDARY OUTCOMES:
Overall Survival under T-DM1 | From study treatment period until death, up to 1 year on average
  The Overall survival (OS) defined from the start of treatment to the date of death from any cause (cohort A) Overall survival (OS) of subjects in cohort A will be analysed as time-to-event study and estimated using Kaplan-Meier method
Duration of Response under T-DM1 | During study treatment period until disease progression or death, up to 1 year on average
  The Duration of response (DoR) defined as the time from the date of first documentation of response (CR or PR) to disease progression or death, in participants who achieve complete or partial response assessed by metabolic response (cohort A) DoR of subjects in cohort A will also be analysed as time-to-event study and estimated using Kaplan-Meier method
Disease Control Rate under T-DM1 | From study treatment period until disease progression or death, up to 1 year on average
  The disease control rate (DCR) defined as absence of disease progression The DCR of subjects in cohort A will be described as proportion with two-sided 95% binomial proportion confidence intervals.
Safety of T-DM1 | From study treatment period until progression disease, start of new anti-cancer treatment or death, up to 1 year on average
  Incidence, nature, and severity of adverse events, including but not limited to drug induced liver injury The intensity of all AEs will be graded according to the NCI-CTCAE version 5.0 on a five-point scale (Grade 1 to 5)

OTHER OUTCOMES:
Correlation between "HER2 positivity" assessments in tumour tissue, HER2-PET/CT and ctDNA | Through study completion, up to 2 years depending on the cohort
  To characterize the correlation between different methods of HER2-expression assessment (i.e., tissue evaluation [immunohistochemistry and in situ hybridization], molecular imaging [HER2-PET/CT], and circulating tumour DNA [ctDNA]) (cohorts A and B)
Correlation between genomic and transcriptomic alterations with best overall response | Through study completion, up to 2 years depending on the cohort

CONTACTS AND LOCATIONS:
Overall Officials: Martine Piccart, Md, PhD, Study Chair — Jules Bordet Institute

IPD SHARING:
Plan to Share IPD: No